CLINICAL TRIAL: NCT01681381
Title: A Prospective, Open Label, Randomized Study to Evaluate Safety And Effectiveness Of The Tivoli® Biodegradable Polymer Rapamycin-Eluting Stent and The FIREBIRD2® Rapamycin-Eluting Coronary CoCr Stent For Treatment Coronary Revascularization
Brief Title: Evaluate Safety And Effectiveness Of The Tivoli® DES and The Firebird2® DES For Treatment Coronary Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Essen Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-LOVE-IT2
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2012-11

CONDITIONS: Ischemic Heart Disease; Myocardial Ischemia; Coronary Artery Lesions,Primary; Coronary Disease; Acute Coronary Syndrome; Furcation Lesion of Coronary Artery
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Firebird2® DES (Active Comparator): Device:Firebird2® DES The Firebird2® rapamycin-eluting stent (Firebird2® DES) is an open cell balloon expandable cobalt chromium stent coated with a biocompatible durable styrene-butylenes-styrene (SBS) polymer containing rapamycin at a dose of 9 micrograms per millimeter of stent length.
  Interventions: Device: Tivoli® DES; Device: Firebird2® DES
- Tivoli® DES (Experimental): Device:Tivoli® DES The Tivoli® DES is an open cell balloon expandable cobalt chromium stent coated with a bio-gradable polymer (PLGA) containing rapamycin at a dose of 8 micrograms per millimeter of stent length.
  Interventions: Device: Tivoli® DES; Device: Firebird2® DES

INTERVENTIONS:
Device: Tivoli® DES — Device:Tivoli® DES The Tivoli® DES drug eluting stent(Tivoli® DES) is an open cell balloon expandable cobalt chromium stent coated with a bio-gradable polymer (PLGA) containing rapamycin at a dose of 8 micrograms per millimeter of stent length. In vitro assays have shown that about 50% of the drug releasing in 1 week and approximately 80% releasing in 28 days. The polymer may be degraded in 3 to 6 months in human body. This stent is supplied pre-mounted on a delivery catheter and is available in the following sizes: lengths of 10、15、18、21、25、30、35 mm and diameters of 2.5、2.75、3.0、3.5、4.0 mm.
Device: Firebird2® DES — The Firebird2® rapamycin-eluting stent (Firebird2® DES) is an open cell balloon expandable cobalt chromium stent coated with a biocompatible durable styrene-butylenes-styrene (SBS) polymer containing rapamycin at a dose of 9 micrograms per millimeter of stent length. In vitro assays have shown that about 50% of the drug elutes in 1 week and approximately 90% elutes in 1 month. This stent is supplied pre-mounted on a delivery catheter and is available in the following sizes: lengths of 13, 18, 23, 29, 33 mm and diameters of 2.25, 2.5, 2.75, 3.0, 3.5, 4.0 mm.

SUMMARY:
This is a prospective, multi-center, open label, randomized study to evaluate the efficacy and safety of The TIVOLI Biodegradable polymer Rapamycin-Eluting Stent comparing with The FIREBIRD2™ Rapamycin-eluting Stent (DES) for Treatment Coronary Revascularization.

ELIGIBILITY:
Inclusion Criteria:

* • The patient must be ≥18 of age;

  * Symptomatic ischemic heart disease and/or objective evidence of myocardial ischemia including chronic stable coronary artery disease, or acute coronary syndrome including non-ST-elevation and ST-elevation myocardial infarction;
  * Acceptable candidate for CABG;
  * The patient is willing to comply with specified follow-up evaluations;4.Patients who agree to accept the follow-up visits.
  * Patients can understand the study objectives psychologically and linguistically and show the sufficient compliance to the study protocol. Patients present acceptance of the risks and benefits described in the informed consent form.

Angiographic Inclusion criteria:

* At least one lesion with a diameter stenosis >70% or more suitable for coronary stent implantation in a vessel with a reference diameter ranging from 2.5 mm to 4.0 mm;
* Patients with multi-lesion or multi-vessel coronary disease, must have successful treatment (<30% diameter stenosis visual estimate) of the first treated lesion prior to treatment of other lesions at the same brand of stent. Staged (planned) procedures must be performed within 30 days of the index procedure.

Exclusion Criteria:

* General Exclusion Criteria

  * Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure.
  * Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated or in which patient will not be able to comply with dual antiplatelet therapy for at least 1 year;
  * Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
  * Left ventricular function <40%;
  * Cardiogenic shock or hemodynamic compromise requiring pressors and/or inotropes or mechanical support;
  * Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, stainless steel alloy, cobalt chromium, Rapamycinry , styrene-butylenes-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately pre-medicated;
  * Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
  * Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.
  * Existing impairment in liver and kidney.
  * Extremely tortuous and/or calcification lesions.

Angiographic exclusion criteria:

• Two or more chronic total occlusions in the proximal half of the epicardial coronary artery which cannot be recannalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2790 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Ischemia-driven Target Lesion Failure (TLF) which is a composite of cardiac death, myocardial infarction (Q and non-Q wave) and target lesion revascularization (TLR) at 12 months post-procedure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Han Yaling, Prof., Principal Investigator — The General Hospital of Shenyang Military Region
Locations (1):
- The General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Han Y, Xu B, Xu K, Guan C, Jing Q, Zheng Q, Li X, Zhao X, Wang H, Zhao X, Li X, Yu P, Zang H, Wang Z, Cao X, Zhang J, Pang W, Li J, Yang Y, Dangas GD. Six Versus 12 Months of Dual Antiplatelet Therapy After Implantation of Biodegradable Polymer Sirolimus-Eluting Stent: Randomized Substudy of the I-LOVE-IT 2 Trial. Circ Cardiovasc Interv. 2016 Feb;9(2):e003145. doi: 10.1161/CIRCINTERVENTIONS.115.003145. PMID 26858080
- [Derived] Han Y, Xu B, Jing Q, Lu S, Yang L, Xu K, Li Y, Li J, Guan C, Kirtane AJ, Yang Y; I-LOVE-IT 2 Investigators. A randomized comparison of novel biodegradable polymer- and durable polymer-coated cobalt-chromium sirolimus-eluting stents. JACC Cardiovasc Interv. 2014 Dec;7(12):1352-60. doi: 10.1016/j.jcin.2014.09.001. Epub 2014 Nov 12. PMID 25440887